CLINICAL TRIAL: NCT02092181
Title: A Pilot Study of Mirabegron and Behavioral Modification Including Pelvic Floor Exercise for Overactive Bladder in Parkinson's Disease. (MAESTRO)
Brief Title: A Pilot Study of Mirabegron and Behavioral Modification Including Pelvic Floor Exercise for Overactive Bladder in Parkinson's Disease (MAESTRO)
Acronym: Maestro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Burdick, MD (Individual)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Burdick, MD, Principal Investigator, Burdick, Daniel, M.D.
Organization: Burdick, Daniel, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DBPA-2013-01
Record Dates: First submitted 2014-03-07; First posted 2014-03-20 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Parkinsons Disease
MeSH Terms: conditions — Parkinson Disease | interventions — mirabegron; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron (Active Comparator): 1:1 randomization to receive Mirabegron 25 mg daily or placebo at visit 2. At visit 3 all subjects who have tolerated Mirabegron 25 mg daily (no adverse events on this dose) will be up-titrated to Mirabegron 50 mg daily. This will be dispensed as two 25mg tablets or, for those in the placebo arm, two placebo tablets.
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): 1:1 randomization to receive Mirabegron 25 mg daily or placebo at visit 2. At visit 3 all subjects who have tolerated Mirabegron 25 md daily (no adverse events on this dose) will be up-titrated to Mirabegron 50 mg daily. This will be dispensed as two 25mg tablets or , for those in the placebo arm, two placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — 25 mg po daily for 32-40 days. Following up-titration to 50 mg po daily. This is pending no adverse events on the 25 mg dose.
  Other Names: Mirabetriq
  Arms: Mirabegron
Drug: Placebo — Placebo 25 mg po daily. Following up-titration to 50 mg po daily. This is pending no adverse events on the 25 mg dose.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the study drug, Mirabegron, is safe and effective in treating symptoms of Overactive Bladder in people with Parkinson's Disease.

DETAILED DESCRIPTION:
This study is a randomized 1:1 placebo-controlled 10-week study of Mirabegron as add-on therapy to an educational intervention of behavioral modification including pelvic floor exercise (PFE) in a cohort of 40 Parkinson's subjects over the age of 30 with overactive bladder (OAB). Active drug will be Mirabegron 25 mg daily with up-titration to 50 mg daily after 5 weeks. Subjects will be enrolled based on response to an overactive bladder questionnaire at visit 2.

Enrolled subjects will have 4 study visits to the clinic as well as 2 phone visits.

Enrolled subjects will be asked to record urinary symptoms and pelvic floor exercises in a diary at 3 separate time points for a 72 hour period.

ELIGIBILITY:
Inclusion Criteria:-

* Diagnosis of Parkinsons by United Kingdom brain bank criteria
* Age > 30 years old
* No change in Parkinsons medications during the 4 weeks preceding screening, with no dose changes during the study, except that PRN (as needed) doses of carbidopa/levodopa will be allowed to address periodic worsening of parkinsonian symptoms.
* Patient willing and able to complete micturition diary
* Urinary urgency (≥ 8 entries of bladder urgency score > 2) in 72hr voiding diary during screening period
* Micturition frequency ≥ 8 / 24hr or incontinence ≥ 2 episodes in 72hr voiding diary during screening period
* Use of other medication that could influence bladder function, other than those specifically prohibited (see below), will be permitted as long as the dose is stable for 4 weeks preceding screening, with no dose changes during the study.
* Patient expects to have valid health insurance for the duration of the study period

Exclusion Criteria:

* Women who are breast-feeding, pregnant or have potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures).
* Cognitive deficits that in the opinion of the investigator would interfere with the subject's ability to give informed consent or perform study testing.
* Screening blood pressure > 165 systolic or 100 diastolic
* Heart rate > 100
* History of allergy to Mirabegron.
* Screening post-void residual > 200ml
* Evidence of urinary tract infection at screening
* History of chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs
* Intravesical botulinum toxin treatment within the previous six months of screening.
* Presence of Interstim device
* Use of indwelling catheter or self-catheterization
* Concurrent use of thioridazine, flecainide, propafenone, or Digoxin
* Concurrent use of warfarin (Coumadin)
* Use of one of the anti-cholinergic bladder medications specified below within 14 days of the screening visit. Subjects who have used one of these medications in the past but discontinued it at least 14 days prior to the screening visit can be enrolled.
* Screening estimated glomerular filtration rate (eGFR) < 60, AST ( aspartate aminotransferase ) or ALT ( alanine aminotransferase ) > 2x upper limit of normal
* Any other serious and/or unstable medical condition
* Participation in other drug studies or use of other investigational drugs within 30 days prior to Screening Visit.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Burdick, MD, Principal Investigator — Evergreen Health; Pinky Agarwal, MD, Principal Investigator — Evergreen Health
Locations (1):
- Evergreenhealth Booth Gardner Parkinsons Care Center, Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who have met exclusion criteria.
Groups:
- Mirabegron; Placebo: 1:1 randomization to receive Mirabegron 25 mg daily or placebo at visit 2. At visit 3 all subjects who have tolerated Mirabegron 25 md daily (no adverse events on this dose) will be up-titrated to Mirabegron 50 mg daily. This will be dispensed as two 25mg tablets or , for those in the placebo arm, two placebo tablets.
  Mirabegron: 25 mg po daily for 32-40 days. Following up-titration to 50 mg po daily. This is pending no adverse events on the 25 mg dose.
  Placebo: Placebo 25 mg po daily. Following up-titration to 50 mg po daily. This is pending no adverse events on the 25 mg dose.
Period: Overall Study
Arm/Group | Mirabegron | Placebo
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Mean (Full Range); unit: years]
  Age,mean | 66 [53 to 85] | 67 [60 to 81] | 67 [53 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Daily Overactive Bladder-Symptom Composite Score.
Description: The primary outcome measure will be the change in the mean daily Overactive Bladder-Symptom Composite Score (OAB-SCS) from baseline (visit 2) to visit 4.
  The Over active Bladder- Symptom Composite Score requires subjects to record the severity of urgency of each micturition over a 72 hour period. Subject ratings ranges from 1 to 6 for each micturition as follows: 1. Not at all, 2.A little bit, 3.Somewhat 4.Quite a bit, 5. A great deal, 6. A very great deal. Maximum score depends on number of micturition episodes in the 72 hour period, as the rating of each episode is summed to get the total score. Higher scores indicate worse symptoms of overactive bladder.
Time Frame: 7-82 days. From visit 2 (baseline) to visit 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -3.2 (8.4) | -8.9 (7.9)

2. Secondary Outcome: Overactive Bladder Questionnaire Symptom Severity Scale( OAB-q)
Description: Overactive Bladder questionnaire symptom severity scale (OAB-q), Visit 3 and Visit 4 vs. baseline Scale ranges from 8 to 48 the higher score indicating worse symptoms.
Time Frame: baseline (7-14 days post visit 1), visit 3( 32-40 days post visit 2) and visit 4(74-82 days post visit 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Week 3/baseline | -4.14 (5.2) | -3.2 (4.8)
  Week4/baseline | -2.6 (7.9) | -8.6 (11.3)

3. Secondary Outcome: Non- Motor Symptoms Scale (NMSS)
Description: Non-Motor Symptoms Scale (NMSS), which includes questions about 9 different categories of non-motor symptoms in PD, including urinary symptoms; Visit 3 and Visit 4 vs. baseline.
  Symptoms assessed over the last month. The scale ranges from 0 to 360, with higher scores indicating worse symptoms.
Time Frame: baseline (7-14 days post visit 1), visit 3 (32-40 days post visit 2) and visit 4 (74-82 days post visit 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  visit 3/baseline | -7.5 (15.4) | -19.6 (18.9)
  visit 4/baseline | -10.5 (18.5) | -17.9 (23)

4. Secondary Outcome: Patient Perception of Bladder Condition
Description: Patient Perception of Bladder Condition at Visit 3 and Visit 4 vs. baseline. the scale ranges from 1 to 6 with higher score indicating worse outcome
Time Frame: baseline (7-14 days post visit 1), visit 3 (32-40 days post visit 2) and visit 4 (74-82 days post visit 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  V3/baseline | -0.35 (2.09) | -0.7 (0.5)
  V4/baseline | -0.38 (1.9) | -1.2 (2.18)

5. Secondary Outcome: Subjects Global Impression of Change
Description: Subject's Global Impression of Change at Visit 3 and Visit 4 vs. baseline the scale ranges from 0 to 7 with higher score indicating worse out come .
Time Frame: baseline (7-14 days post visit 1), visit 3 (32-40 days post visit 2) and visit 4 (74-82 days post visit 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  visit 3/baseline | 3.5 (1.8) | 3.0 (1.3)
  visit 4/baseline | 3.5 (2.2) | 2.6 (1.1)

6. Other Pre Specified Outcome: Change in Mean Daily OAB-SCS Visit 3 vs Baseline
Description: as for outcome 1
Time Frame: baseline (7-14 days post visit 1) and visit 3 (32-40 days post visit 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  visit 3 (32-40 days post visit 2 | 3.5 (1.8) | 3.07 (1.3)
  baseline (7-14 days post visit 1) | 3.5 (2.2) | 2.6 (1.2)

7. Other Pre Specified Outcome: Change in Mean Number of Incontinence Episodes Per 24 Hours
Description: Subjects recorded in a 72-hour micturition diary the number of episodes of urinary incontinence, and this is averaged per 24 hours. Higher scores indicate more episodes of incontinence and thus worse outcome.
Time Frame: baseline vs visit 3 (32-40 days post baseline) and baseline vs. visit 4 ((74-82 days post visit 2)
Measure: Mean (Standard Deviation); unit: episodes per 24 hrs
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 15 | 15
episodes per 24 hrs
  V3 vs baseline | -0.06 (0.82) | -0.11 (1.0)
  V4/baseline | 0.12 (1.24) | -0.61 (1.9)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Mirabegron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 9/15 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=15) | Placebo (N=15)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=15) | Placebo (N=15)
Extreme Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Cold symptons (Infections and infestations) | 0 (0) | 2 (2)
Falls (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Hallucinations (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
itchy/swollenhands (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sinus infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
foot or knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Vascular disorders) | 1 (1) | 0 (0)
edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
Sore throat (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
loose stools (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartbun (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-04-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT02092181/Prot_000.pdf